CLINICAL TRIAL: NCT01586169
Title: A Pharmacovigilance Study on the Safety of Integrated Treatment of Trachoma and Lymphatic Filariasis in Children and Adults Living in the Sikasso Region of Mali
Brief Title: Safety of the Co-administration of Three Drugs for Trachoma and Lymphatic Filariasis Elimination
Acronym: AZIVAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Appui à la lutte contre la Maladie (Other)
Collaborators: International Trachoma Initiative (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNAM/AZIVAL/01; 0958/FMPOS (Other: FMPOS)
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Parasitic Diseases; Bacterial Diseases
Keywords: Albendazole; Ivermectin; Azithromycin; Lymphatic filariasis; Trachoma; Safety
MeSH Terms: conditions — Parasitic Diseases; Bacterial Infections; Elephantiasis, Filarial; Trachoma | interventions — Ivermectin; Azithromycin; Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: triple co administration at once of the combination of Albendazole + ivermectin + azithromycin — Albendazole 400mg + ivermectin according to the height + azithromycin according to the height at once
  Other Names: Albendazole; Mectizan; Zithromax

SUMMARY:
The purpose of this study is to determine whether the triple co administration of albendazole, ivermectin and azithromycine is as safe as the current treatment scheme that consists to treat with albendazole plus ivermectin together and a week later to treat with azithromycin in areas co endemic for lymphatic filariasis and trachoma.

DETAILED DESCRIPTION:
Infectious diseases such as trachoma and lymphatic filariasis are public health problems in regions of Africa and Asia. Elimination programs exist for the two diseases, and their treatment by different groups of health workers is both costly and inefficient.

Thus, a study evaluating the safety and feasibility of an integrated mass treatment of trachoma and lymphatic filariasis with azithromycin associated with albendazole and ivermectin was instituted in 4 villages of the region of Sikasso in Mali (West Africa) co endemic for lymphatic filariasis and trachoma.

It was an open label randomized clusters type on the assessment of the safety of the triple co administration of azithromycin, ivermectin and albendazole (experimental regimen) as compared to the administration of the co administration of albendazole plus ivermectin followed by the that of azithromycin a week later (current standard recommended regimen) within subjects of 5 to 65 years old, willing and able to swallow the study drugs.

Clinical evaluation of adverse events in all study participants was done on day 0, day 8, and day 15 after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have been residing in the village for at least three months;
* Must be 90 cm tall or more;
* Must be between 5 years and 65 years of age;
* Must not be pregnant;
* Must not be lactating.

Exclusion Criteria:

* Subjects under 5 years of age or less than 90 cm in height;
* Subjects over 65 years of age;
* Subjects who cannot swallow tablets;
* Subjects who are sick and bedridden;
* Pregnant women (clinical appreciation in the study);
* Lactating women;
* History of allergies to the drugs being studied (azithromycin, ivermectin, albendazole).

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Establish the incidence of adverse events associated with the mass triple drug administration | From Day 0 to Day 15 post treatment

SECONDARY OUTCOMES:
Establish the incidence of serious adverse events associated with the mass triple drug administration | From Day 0 to Day 15 post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Samba O Sow, MD, MPH, Principal Investigator — CNAM, Mali
Locations (1):
- Centre National D'Appui a la lutte contre la Maladie, Bamako, Mali, Mali

REFERENCES:
- [Derived] Coulibaly YI, Dicko I, Keita M, Keita MM, Doumbia M, Daou A, Haidara FC, Sankare MH, Horton J, Whately-Smith C, Sow SO. A cluster randomized study of the safety of integrated treatment of trachoma and lymphatic filariasis in children and adults in Sikasso, Mali. PLoS Negl Trop Dis. 2013 May 9;7(5):e2221. doi: 10.1371/journal.pntd.0002221. Print 2013. PMID 23675549